CLINICAL TRIAL: NCT00337701
Title: Biojector 2000 Open-Label Safety Study (BOSS) to Evaluate Signs and Symptoms Associated With a Needle-free Injection Device for Administration of Fuzeon to Patients With HIV-1 Infection
Brief Title: BOSS Study: A Study of Fuzeon Using the Needle-Free Biojector 2000 in Patients With HIV-1 Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Trimeris (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML19849
Record Dates: First submitted 2006-06-15; First posted 2006-06-16 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: enfuvirtide [Fuzeon]
- 2 (Experimental)
  Interventions: Drug: enfuvirtide [Fuzeon]

INTERVENTIONS:
Drug: enfuvirtide [Fuzeon] — 90mg sc bid by Biojector 2000 NFID for 8 weeks
  Arms: 1
Drug: enfuvirtide [Fuzeon] — 90mg sc bid by standard needle and syringe for 4 weeks, followed by 90mg sc bid by Biojector 2000 NFID for 4 weeks.
  Arms: 2

SUMMARY:
This study will evaluate the signs and symptoms associated with Fuzeon injection (90mg sc) using the B2000 needle-free injection device, in HIV-1 positive patients experienced to Fuzeon treatment, but having difficulty tolerating long-term (>4 weeks) administration of Fuzeon with the standard needle and syringe. Patients will be randomized to the B2000 device or the standard needle and syringe for 4 weeks; all patients will use the B2000 device for the next 4 weeks. The anticipated time on study treatment is <3 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=16 years of age;
* current or former Fuzeon user who may benefit from needle-free administration of Fuzeon;
* naive to use of the B2000 device;
* positive test results for human immunodeficiency virus infection.

Exclusion Criteria:

* patients naive to Fuzeon;
* inability to self-inject Fuzeon, or no reliable caregiver to administer injections;
* evidence of active, untreated, opportunistic infections.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2006-06; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Composite endpoint (pain, induration, nodules/cysts) | Throughout study

SECONDARY OUTCOMES:
AEs and ISRs | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (40):
- United States (38):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Fountain Valley, California
  - Hayward, California
  - Long Beach, California
  - Los Angeles, California
  - Palm Springs, California
  - San Francisco, California
  - Santa Clara, California
  - Denver, Colorado
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - North Miami Beach, Florida
  - Orlando, Florida
  - Plantation, Florida
  - Port Saint Lucie, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Baltimore, Maryland
  - Silver Spring, Maryland
  - Boston, Massachusetts
  - Berkley, Michigan
  - St Louis, Missouri
  - Somers Point, New Jersey
  - Voorhees Township, New Jersey
  - New York, New York
  - Rochester, New York
  - Winston-Salem, North Carolina
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Fort Worth, Texas
  - Galveston, Texas
  - Houston, Texas
  - Hampton, Virginia
  - Spokane, Washington
- Puerto Rico (2):
  - Ponce
  - Santurce